CLINICAL TRIAL: NCT03094780
Title: A Structured Multidisciplinary Quality of Life Intervention for Patients Receiving Radiation Therapy for Advanced Cancer Treatment & Their Caregivers: A Telemedicine Project
Brief Title: Quality of Life Intervention for Patients Receiving Radiation Therapy for Advanced Cancer Treatment and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew M. Clark, Ph.D., L.P., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-009226
Record Dates: First submitted 2016-08-23; First posted 2017-03-29 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Quality of Life; Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quality of Life Counseling (Other)
  Interventions: Behavioral: Quality of life counseling; Other: Video-conference quality of life counseling

INTERVENTIONS:
Behavioral: Quality of life counseling — Will receive quality of life counseling from PI, social workers, and physical therapists
Other: Video-conference quality of life counseling — Participants may video-conference to other sites to participate in group session dependent on Florida, Northfield and Arizona enrollment

SUMMARY:
This study will use video technology in conjunction with in-person participation. This is a pilot project, where all enrolled participants will receive the multidisciplinary intervention. Participants (patients and caregivers) from Mayo Clinic Rochester will attend an in-person group session, and participants (patients and caregivers) from Mayo Clinic Florida or Northfield Mayo Clinic Radiation Oncology Center will participate through the use of video conferencing. The goals are to examine feasibility (percent of eligible patients and caregivers who enroll), attrition, and adherence (attend at least four of the six sessions), to determine any differences between the two formats, and to examine potential QOL differences as a result of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age.
* Ability to attend all treatment sessions and follow-up.
* Ability to provide written informed consent.
* Ability to participate in all aspects of the study.
* Initial diagnosis of cancer must have been 12 months prior to study entry.
* Intermediate to poor prognosis, defined as an expected 5-year survival of 0%-50% in the judgment of the physicians entering the patient on the study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1, or 2.
* 1 week of planned cancer treatment (radiation or chemotherapy) at Mayo Clinic.
* Has a caregiver also willing to participate.
* Willingness to get e-mail/text reminder to complete the follow-up survey or complete the follow-up survey with a study coordinator by phone.

Exclusion Criteria:

* Expected survival of <6 months.
* Active substance abuse (alcohol or drug).
* Participation in other psycho-social research trials.
* Active untreated thought disorder (bipolar illness, schizophrenia, etc.).
* Untreated suicidal intent or plan.
* In need of psychiatric hospitalization.
* Recurrent disease after disease-free interval of >6 months.
* Previous cancer 5 years (except non-melanoma skin cancer and/or second cancer diagnosed at approximately the same time as this cancer).
* Use of Proton Beam Radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2018-12 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Change in the participant's QOL at 4 weeks (end of the intervention) | baseline, 4 weeks
  Quality of Life, 0 to 10. 7 or higher is positive.
Change in the participant's QOL at 26 weeks | baseline, 26 weeks
  Quality of Life, 0 to 10. 7 or higher is positive.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Clark, Ph.D., L.P., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Northfield, Minnesota
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials